CLINICAL TRIAL: NCT02109861
Title: Phase 0 Microdose Study to Evaluate the Effect of Melphalan, Bortezomib and Dexamethasone on Cellular Gene-expression in Patients With Multiple Myeloma
Brief Title: Microdose Study of Melphalan, Bortezomib and Dexamethasone
Acronym: Phase-0-MM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henrik Gregersen (Other)
Responsible Party: Sponsor-Investigator, Henrik Gregersen, Consultant haematologist, MD, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KFE2011.06; 2011-003791-37 (EudraCT Number)
Record Dates: First submitted 2014-01-15; First posted 2014-04-10 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Phase 0 study; Microdose study; Micro array; Gene expression profiling
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Melphalan (Experimental): A microdose of 2 mg/m2 iv Melphalan (1% of standard dose) is given two hours prior to planned standard dose Melphalan
  Interventions: Drug: Melphalan
- Bortezomib (Experimental): A microdose of 0.013 mg/m2 iv Bortezomib (1% of standard dose) is given two hours prior to planned standard dose Bortezomib
  Interventions: Drug: Bortezomib
- Dexamethasone (Experimental): A microdose of 0.4 mg iv Dexamethasone (1% of standard dose) is given two hours prior to planned standard dose of Dexamethasone
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Melphalan — A microdose of 2 mg/m2 iv Melphalan (1% of standard dose) is given two hours prior to planned standard dose Melphalan
  Other Names: Alkeran®
  Arms: Melphalan
Drug: Bortezomib — A microdose of 0.013 mg/m2 iv Bortezomib (1% of standard dose) is given two hours prior to planned standard dose Bortezomib
  Other Names: Velcade®
  Arms: Bortezomib
Drug: Dexamethasone — A microdose of 0.4 mg iv Dexamethasone (1% of standard dose) is given two hours prior to planned standard dose of Dexamethasone
  Other Names: Dexaven®)
  Arms: Dexamethasone

SUMMARY:
The purpose of the study is to identify specific genes that are up- or downregulated in multiple myeloma patients who receive a microdose of either Melphalan (Alkeran®), Bortezomib (Velcade®) or Dexamethasone (Dexaven®). The study treatment constitutes 1% of the planned standard myeloma treatment and will be given two hours prior to standard treatment. Blood samples are taken at baseline, 15, 30, 60 and 120 minutes for microarray analysis.

ELIGIBILITY:
Inclusion Criteria:

* Planned treatment for Multiple Myeloma (newly diagnosed as well as relapse and refractory disease) with one of the following chemotherapy regimens: 1) Highdose melphalan, 2) Bortezomib or 3) Dexamethasone
* 18 years or older.
* Understand and have the will to sign the informed consent.

Exclusion Criteria:

* Prior treatment with the study drug
* Received treatment with biphosphonates in the week prior to study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in gene expression at 15, 30, 60, 120 minutes upon microdose drug exposure. | Prior to microdose and 15, 30, 60 and 120 minutes post-microdose
  The primary outcome measure is determination of differential and significantly expressed genes across time successive samples from each individual patient. The analysis will be based on global gene expression profiling and differentially expressed genes will be identified using pairwise comparisons of samples means by two sample t-tests and corrections for multiple testing.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Gregersen, MD, PhD, Principal Investigator — Aalborg University Hospital, Department of Haematology, 9000 Aalborg, Denmark
Locations (1):
- Department of Haematology, Aalborg University Hospital, Aalborg, Denmark